CLINICAL TRIAL: NCT00137033
Title: A Multicenter, Randomized, Active-Controlled Comparison Study of the Incidence of Gastroduodenal Ulcers Associated With Celecoxib and Low Dose ASA Versus Naproxen and Low Dose ASA in Healthy Subjects (50-75 Years of Age)
Brief Title: Celebrex Low Dose ASA Study Examining the Incidence of Gastroduodenal Ulcers in a Healthy Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A3191171
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Peptic Ulcers
MeSH Terms: conditions — Peptic Ulcer | interventions — Celecoxib; Naproxen

INTERVENTIONS:
Drug: Celecoxib
Drug: Naproxen
Drug: ASA

SUMMARY:
The aim of the current study is to replicate the COXA-0508-258 study in a multicenter, US setting, using a lower dose of ASA. It is expected that this study will not only confirm the results of the 258 study but show that the incidence of UGI ulcers on celecoxib is significantly less than on traditional NSAIDs and the incidence of UGI ulcers on celecoxib increases with the addition of ASA, but still is lower than traditional NSAIDs plus/minus ASA. This 7-day study is designed to compare the incidence of gastroduodenal ulcers associated with celecoxib 200 mg QD and low dose aspirin 81 mg QD and with naproxen 500 mg BID plus low dose aspirin 81 mg QD in healthy adults(50-75 years of age).

ELIGIBILITY:
Inclusion Criteria:

* A healthy adult between 50 and 75 years of age inclusive: of normal clinical laboratory test results during the Screening Visit or, if abnormal, are not clinically significant in the Investigator's opinion.

Exclusion Criteria:

* A gastric, pyloric channel or duodenal ulcer (defined as any break in the mucosa at least 3 mm in diameter with unequivocal depth) or more than 5 erosions in the stomach or duodenum ( the UGI endoscopic score greater or less) on the baseline UGI endoscopy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 605
Dates: Start 2004-09; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Compare the incidence of gastroduodenal endoscopic ulcers between celecoxib 200 mg QD plus ASA 81 mg QD vs. naproxen 500 mg BID plus ASA 81 mg QD in healthy subjects (50-75 years old).

SECONDARY OUTCOMES:
Compare the incidence of gastroduodenal endoscopic ulcers between celecoxib plus ASA vs placebo plus ASA in healthy subjects (50-75 years of age) Compare the incidence of gastroduodenal endoscopic ulcers between naproxen plus ASA vs. placebo plus ASA

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocoee, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Davenport, Iowa
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Chevy Chase, Maryland
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Chesapeake, Virginia